CLINICAL TRIAL: NCT05519735
Title: Multimodal Characterization of Lymphatic Organs and Myocardium in Patients After Acute Myocardial Infarction
Brief Title: Lymphatic Organs and Myocardium After Myocardial Infarction
Acronym: LOMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Theresa Reiter, Principal Investigator, Wuerzburg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 192/21
Record Dates: First submitted 2022-08-22; First posted 2022-08-29 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Myocardial Infarction; Myocardial Injury; Myocardial Inflammation
Keywords: CXCR4; CMR; Lymphatic organs; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; Myocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal imaging (Other): Multimodal imaging approach. This includes a CXCR4 targeted PET/CT ([68Ga]Pentixafor) during the acute hospital stay, and serial CMR and Echo imaging.
  Interventions: Diagnostic Test: Multimodality Imaging

INTERVENTIONS:
Diagnostic Test: Multimodality Imaging — Patients receive CXCR4-targeted PET/CT, CMR and Echo

SUMMARY:
The adaptive immune response plays an important role in myocardial healing and remodeling after acute myocardial infarction in patients. Therefore, the involved lymphocytes represent a novel target for therapeutic interventions. However, there are no established blood-derived biomarkers to predict the quantity and quality of the adaptive immune response to cardiac injury. Multimodal imaging of the heart and immunologic organs might provide such information.

Recent retrospective analysis of patients after MI revealed enlarged mediastinal lymph nodes associated with increased CXCR4 radiotracer accumulation, thereby indicating that CXCR4 PET-based lymph node imaging provides a non-invasive quantitative readout of the local adaptive immune response. These considerations are further fuelled by the fact that, within lymph nodes, CXCR4 is expressed almost exclusively on lymphocytes, whereas various other cell types express CXCR4 within the myocardium.

This leads to the hypothesis that the size of mediastinal lymph nodes and their respective CXCR4 PET signals correlate with the adaptive immune response to cardiac injury and might provide predictive information for functional cardiac decline during follow-up.

This prospective clinical study will use multimodal imaging to monitor chemokine receptor 4 (CXCR4) expression in the lymph nodes, myocardium, spleen, and bone marrow after acute MI. The combination of cardiac magnetic resonance (CMR), echocardiography, and positron emission tomography (PET) along with blood collection for immunophenotyping will allow to determine i) if the size of mediastinal lymph nodes and their respective PET-derived CXCR4 signals at baseline correlate with the adaptive immune response to acute cardiac injury; and ii) if they predict cardiac adverse remodelling during longitudinal follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute myocardial infarction (STEMI) who were treated with immediate catheterization
* stable clinical course
* male/female, above 18 years old

Exclusion Criteria:

* hemodynamic instablity > 48 h after immediate catherization
* known CAD
* known structural heart disease
* multi vessel disease
* NSTEMI
* sarcoidosis
* immunosuppressive therapy
* acute inflammatory disease
* no consent obtainable
* contraindiations for CMR
* impaired renal function
* active cardiac implants, ferromagnetic implants
* pregnancy, breast-feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
CXCR4 PET-derived uptake after myocardial infarction | 12 months
  Semi-quantitative assessment of CXCR4-derived radiotracer accumulation in the myocardium, mediastinal lymph nodes, bone marrow and spleen in patients after myocardial infarction. For quantitative analysis, standardized uptake values (SUV) will be calculated in organs of interest.

SECONDARY OUTCOMES:
Correlation of quantitative parameters (SUV) with peripheral lymphocytes | 12 months
  SUV of organs of interest are correlated to the phenotype of peripheral lymphocytes in the peripheral blood after myocardial infarction.
Time course of SUV after myocardial infarction | 12 months
  PET/CT scans for each patient will be allocated to either day 3-4 or day 5-8 after myocardial infarction. SUV of organs of interest will be correlated to time point of imaging.
Correlation of myocardial damage to SUV | 12 months
  CMR will determine the extend of myocardial damage as necrotic volume, volume of MVO and myocardial edema. These findings will be correlated to SUV.
Correlation of SUV with the clincial course | 12 months
  Myocardial function (LVEF) and scar volumes as determined by CMR will be correlated to the intital SUV in order to correlate the clinical outcome to the tracer activity.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Reiter, MD, Principal Investigator — Wuerzburg University Hospital; Rudolf Werner, MD, Principal Investigator — Wuerzburg University Hospital
Locations (2):
- Germany (2):
  - Klinikum Würzburg Mitte, Medizinische Klinik, Würzburg
  - University Hospital Wuerzburg, Würzburg